CLINICAL TRIAL: NCT05441371
Title: Antibacterial Effect of Paradontax Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Odd Carsten Koldsland, Associate professor, University of Oslo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REK 370116
Record Dates: First submitted 2022-06-09; First posted 2022-07-01 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Plaque Induced Gingivitis; Plaque, Dental
Keywords: split mouth; chemical plaque control
MeSH Terms: conditions — Dental Plaque | interventions — Toothpastes

STUDY DESIGN:
Intervention Model Description: Split mouth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test; Parodontax toothpaste (Experimental): 1.st quadrant of subject
  Interventions: Other: Toothpaste; Paradontax
- Control; Regular toothpaste (Placebo Comparator): 2.nd quadrant of subject
  Interventions: Other: Toothpaste; Paradontax

INTERVENTIONS:
Other: Toothpaste; Paradontax — Comparison of Paradontax toothpaste anti-plaque abality versus regular toothpaste

SUMMARY:
The purpose of the study is to test the antibacterial effect of Parodontax toothpaste on plaque formation, and thus gingivitis compared to placebo toothpaste.

Each subject will be given 2 plastic splints that are individually adapted to their quadrant 1 and 2. In the splint in the 1st quadrant, Parodontax test toothpaste will be placed, while in the splint in the 2nd quadrant, regular toothpaste will be placed, which the subject uses daily. Each person's set of teeth is otherwise professionally cleaned.

DETAILED DESCRIPTION:
Each subject will be given 2 plastic splints that are individually adapted to their quadrant 1 and 2. In the splint in the 1st quadrant, Parodontax test toothpaste will be placed, while in the splint in the 2nd quadrant, regular toothpaste will be placed, which the subject uses daily. Each person's teeth is otherwise professionally cleaned.

Home procedure: The subject first rinses the mouth with water for 30 sec. Then both splints are placed on the teeth in the 1st quadrant and 2nd quadrant, respectively, and the rest (lower jaw) is brushed with the subject's regular toothpaste. The brace should be on for 1 min while cleaning the teeth in the lower jaw as usual, with its usual commercial toothpaste. After 1 minute, rinse your mouth with water for 30 seconds. Then the splints are removed and the mouth is immediately rinsed with water for another 30 sec. The procedure is repeated twice a day (morning and evening) for 3 weeks (21 days). In this way, the test person becomes his own control (1st quadrant versus 2nd quadrant), and the individual plaque quality is subordinate to what it would not otherwise be in a 2-group study. Furthermore, individual brushing technique will not be an issue, as we only test the antibacterial effect of the toothpaste in the splint quadrants. It is the antibacterial effect of Parodontax we test, not affected by brushing technique.

Health information that includes age, medication use, allergies, diseases, and tobacco use. Following the test period, registration of plaque (Silness&Loe/Quigley&Hines) and gingival bleeding (Loe&Silness) will be registered

ELIGIBILITY:
Inclusion Criteria:

Healthy people of both sexes

* age 18-35 years
* Have at least three of the following teeth: 16, 15, 14, 13, 23, 24, 25, 26 with healthy gingiva.
* Non-smokers
* Has signed an informed consent document

Exclusion Criteria:

Pregnancy and breast-feeding.

* Any chronic disease Clinical or other symptoms of oral disease
* Any prescribed or over-the-counter systemic or topical medication with the exception of oral contraceptives used within one week prior to the start of the study.
* Haematological and clinical / chemical parameters considered unacceptable by the project manager.
* Use of antibiotics within the last three months before the start of the study.
* Alcohol or drug / drug abuse
* Participation in other clinical studies in the last 4 weeks before the start of the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Plaque Index (PI) | 21 days
  Amount of plaque at surfaces

SECONDARY OUTCOMES:
Gingival bleeding (GI) | 21 days
  Inflammation/bleeding on gentle probing of gingiva
Presence of plaque at entire tooth | 21 days
  Amount of surface covered by plaque visualized by discolouration

CONTACTS AND LOCATIONS:
Overall Officials: Carl Hjortsjø, Ph.D, Study Chair — Head of Institute
Locations (1):
- Dental faculty, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abrahamsen S, Koldsland OC, Preus HR. The anti-plaque effect of high concentration sodium bicarbonate dentifrice on plaque formation and gingival inflammation, irrespective to individual polishing technique and plaque quality. BMC Oral Health. 2023 May 11;23(1):281. doi: 10.1186/s12903-023-03005-y. PMID 37170260